CLINICAL TRIAL: NCT03132220
Title: A Mindfulness Based Cognitive Therapy (MBCT) Resiliency Program for Critical Care Nurses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-0279
Record Dates: First submitted 2017-04-21; First posted 2017-04-27 (Actual); Results first posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-11

CONDITIONS: Burn-Out Syndrome; Work-Related Stress Disorder
Keywords: critical care nurses; mindfulness-based cognitive therapy; Burn-out Syndrome; Post-traumatic Stress Disorder; Cognitive Behavioral Therapy
MeSH Terms: conditions — Burnout, Psychological; Stress Disorders, Post-Traumatic | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Book Club Active Control (Active Comparator): The subject will participate in 16 in-person hours that are broken into sessions for the book club active control intervention. This club will be facilitated by 1-2 instructors. The club will be described as a "fun activity to do outside of work to help reduce work-related stress." The club will be structured similarly to the intervention with respect to time, and homework expectations. Nurses will be prohibited from talking about work stress.
  Interventions: Behavioral: Book Club Active Control Intervention
- MBCT Intervention (Experimental): The subject will participate in 16 in-person hours that are broken into sessions for the Mindfulness-Based Cognitive Therapy intervention. The intervention will be facilitated by 1-2 instructors who are trained in clinical psychology/ social work and are also trained in MBCT. This intervention will include mindfulness activities, didactic learning, homework assignments and group dialogue. This adapted MBCT intervention will follow the empirically-based MBCT intervention for depression structure with fidelity.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy — Mindfulness-Based Cognitive therapy is a 16 in-person hours intervention. The intervention in this population is designed to reduce symptoms of PTSD and BOS and increase resiliency scores.
  Arms: MBCT Intervention
Behavioral: Book Club Active Control Intervention — Participants randomized to the book club active control intervention will meet for 16 in-person hours that are broken into sessions. Books will be assigned to read during homework time and discussions regarding the books will occur during the sessions. The time involved will be similar to the MBCT intervention.
  Arms: Book Club Active Control

SUMMARY:
Developed over 10 years ago, Mindfulness Based Cognitive Therapy (MBCT) synergistically combines mindfulness training and cognitive behavioral therapy and can increase resiliency. In this study, the investigators proposed two aims: Aim #1: To adapt and optimize a MBCT resiliency program specifically for ICU nurses. For this aim, the investigators will engage multiple stakeholder groups to assist the protocol adaptation. Aim # 2: To conduct a pilot clinical trial to determine acceptability of the MBCT resiliency program and the control intervention. In this aim, the investigators will also identify the most feasible randomization level to minimize contamination between the control and intervention groups. Collectively, this proposal will pave the way for a properly designed large multi-center trial of a MBCT resiliency program (MBCT-ICU) to determine its ability to decrease BOS symptoms; and allow nurses to more effectively care for patients in the challenging ICU environment.

DETAILED DESCRIPTION:
The Intensive Care Unit (ICU) is a stressful environment for all critical care healthcare providers. In the United States, there are more than 500,000 critical care (ICU) nurses that treat the most seriously ill patients. These ICU nurses have especially challenging and sometimes overwhelming jobs due to high patient mortality and morbidity, and frequent encounters with ethical dilemmas. The repetitive exposure to these extreme stressors and the inability to adjust to their difficult work environment may cause significant psychological stress. The investigator's multidisciplinary research team was one of the first to identify that ICU nurses have significantly high rates of psychological distress including: symptoms of anxiety and depression, posttraumatic stress disorder (PTSD) and burnout syndrome (BOS).

Work-induced distress initiates a negative cycle that contributes to the unacceptably high ICU nursing turnover rate. Nationally, nursing turnover rates range between 17-20% per year. In the ICU, the growing nursing shortage is particularly concerning. Presently, there are no interventions to reduce BOS in ICU nurses. Many stresses on ICU nurses are inherent to the critical care environment such as performing cardiopulmonary resuscitation and the death of a patient. Therefore, the investigators multidisciplinary research group has focused on enhancing the ability of ICU nurses to adapt to their work environment.

Resiliency enables one to thrive in the face of adversity. Humans respond to stress and trauma in a variety of ways. Some people are resilient; defined as the ability to succeed, to live, and to develop in a positive way despite the stress or adversity that would normally involve the real possibility of a negative outcome. In practice, resilient individuals believe that what they do can have a positive impact on a situation, that some components of the 'system' can be controlled or influenced by one's own actions, that persistent effort is worthwhile, and that setbacks or potentially threatening events are inevitable and surmountable. A variety of qualities are associated with resiliency including the ability to engage the support of others, the belief that stress can be strengthening, and overall optimism. Though some individuals are inherently resilient; resiliency can be learned. Developing resiliency may be one strategy to prevent and treat symptoms of BOS. The investigators have demonstrated that resilient ICU nurses were less likely to have symptoms of anxiety, depression, PTSD, and BOS. The investigators also identified methods used by ICU nurses to promote resiliency and emotional wellness. The investigators ICU nursing pilot program also increased resiliency and decreased symptoms of BOS.

From the investigators prior studies, mindfulness-based stress reduction (MBSR) and cognitive behavioral therapy (CBT) are two modalities currently used by resilient ICU nurses. In the investigators most recent national survey, ICU nurses were eager to learn MBSR and CBT techniques to help reduce symptoms of BOS. Mindfulness Based Cognitive Therapy (MBCT) combines the best of MBSR and CBT, and may build resiliency and reduce BOS symptoms. MBCT was developed by integrating the framework and practices of MBSR and CBT. Classically incorporated into an 8 week course, MBCT uses mindfulness skills to help individuals become aware of negative thoughts and feelings that are activated by stress. MBCT also incorporates CBT techniques to develop a different relationship to those thoughts and feelings, and interrupt the negative thought patterns.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 years or older
2. Employed as a critical care nurse and work at least 20 hours per week as an ICU
3. Baseline score of < 82 on the Connor-Davidson Resilience Scale (CD-RISC)
4. Positive symptoms of at least one BOS dimension using the Maslach Burnout Inventory (MBI):

   * emotional exhaustion score of >17,
   * depersonalization score of >7, or
   * a personal accomplishment score of < 31.

Exclusion Criteria:

1. A self-reported diagnosis of:

   * bipolar or psychotic disorder,
   * active substance dependence, or
   * immediate risk of self-harm or need for hospitalization
2. Unwillingness to participate in the entire study protocol
3. Employment on a time limited contract (i.e. a traveling nurse)

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2019-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Mealer, PhD, Principal Investigator — University of Colorado, Denver; Marc Moss, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
The plan to share IPD is through a limited summary of the data. The information will be de-identified.

RESULTS

PARTICIPANT FLOW:
Groups:
- MBCT Intervention: The subject will participate in 16 hours that are broken into sessions for the Mindfulness-Based Cognitive Therapy intervention. The intervention will be facilitated by 1-2 instructors who are trained in clinical psychology/ social work and are also trained in MBCT. This intervention will include mindfulness activities, didactic learning, homework assignments and group dialogue. This adapted MBCT intervention will follow the empirically-based MBCT intervention for depression structure with fidelity.
  Mindfulness-Based Cognitive Therapy: Mindfulness-Based Cognitive therapy is a 16 hours intervention. The intervention in this population is designed to reduce symptoms of post-traumatic stress disorder (PTSD) and burnout syndrome (BOS) and increase resiliency scores.
- Book Club Active Control: The subject will participate in 16 hours that are broken into sessions for the book club active control intervention. This club will be facilitated by 1-2 instructors. The club will be described as a "fun activity to do outside of work to help reduce work-related stress." The club will be structured similarly to the intervention with respect to time, and homework expectations. Nurses will be prohibited from talking about work stress.
  Book Club Active Control Intervention: Participants randomized to the book club active control intervention will meet for 16 hours that are broken into sessions. Books will be assigned to read during homework time and discussions regarding the books will occur during the sessions. The time involved will be similar to the MBCT intervention.
Period: Overall Study
Arm/Group | MBCT Intervention | Book Club Active Control
Started | 65 | 66
Began Study Sessions | 48 (65 participants randomized to intervention arm;17 lost to f/u prior to study start;48 began sessions) | 58 (66 participants randomized to control arm;8 were lost to f/u prior to study start; 58 began sessions)
Completed | 47 | 54
Not Completed | 18 | 12
Not completed — Lost to Follow-up | 17 | 8
Not completed — Withdrawal by Subject | 1 | 4

BASELINE CHARACTERISTICS:
Population: Baseline demographic data was only captured for the 106 participants who began study sessions.
Groups:
- MBCT Intervention: The subject will participate in 16 hours that are broken into sessions for the Mindfulness-Based Cognitive Therapy intervention. The intervention will be facilitated by 1-2 instructors who are trained in clinical psychology/ social work and are also trained in MBCT. This intervention will include mindfulness activities, didactic learning, homework assignments and group dialogue. This adapted MBCT intervention will follow the empirically-based MBCT intervention for depression structure with fidelity.
  Mindfulness-Based Cognitive Therapy: Mindfulness-Based Cognitive therapy is a 16 hours intervention. The intervention in this population is designed to reduce symptoms of PTSD and BOS and increase resiliency scores.
- Total: Total of all reporting groups
Arm/Group | Book Club Active Control | MBCT Intervention | Total
Number analyzed (Participants) | 58 | 48 | 106
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.4 (7.35) | 33.0 (6.50) | 32.6 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 45 | 99
  Male | 4 | 3 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  % Caucasian | 55 | 44 | 99
  Hispanic, % yes | 2 | 1 | 3
Years practicing as nurse [Mean (Standard Deviation); unit: years] | 6.8 (.91) | 6.5 (.95) | 6.6 (6.7)
Years practicing in Intensive Care Unit (ICU) [Mean (Standard Deviation); unit: years] | 5.3 (.78) | 5.2 (5.9) | 5.3 (5.8)
Medication for anxiety, yes [Count of Participants; unit: Participants] | 8 | 2 | 10
Medication for depression, yes [Count of Participants; unit: Participants] | 11 | 3 | 14
Exercise, yes [Count of Participants; unit: Participants] | 52 | 45 | 97
Practice mindfulness, yes [Count of Participants; unit: Participants] | 14 | 4 | 18
Current therapy/counseling, yes [Count of Participants; unit: Participants] | 12 | 10 | 22
Hospital Anxiety and Depression Scale (HADS)-Anxiety, % positive [Count of Participants; unit: Participants] — The Hospital Anxiety and Depression Scale (HADS) is a 14-item screening scale developed to indicate the possible presence of anxiety and depression3. HADS consists of a 7-item anxiety subscale and a 7-item depression subscale. A score of >8 identifies a positive history of anxiety or depression symptoms 129. The validity of the HADS has been extensively studied in a variety of populations including the general population, general practice and psychiatric population.
  Participants | 45 | 29 | 74
Hospital Anxiety and Depression Scale (HADS)-Depression, % positive [Count of Participants; unit: Participants] — The Hospital Anxiety and Depression Scale (HADS) is a 14-item screening scale developed to indicate the possible presence of anxiety and depression3. HADS consists of a 7-item anxiety subscale and a 7-item depression subscale. A score of >8 identifies a positive history of anxiety or depression symptoms 129. The validity of the HADS has been extensively studied in a variety of populations including the general population, general practice and psychiatric population.
  Participants | 17 | 11 | 28
Maslach Burnout Inventory (MBI)-Emotion Exhaustion, % positive [Count of Participants; unit: Participants] — Maslach Burnout Inventory (MBI) is a 22-item self-report questionnaire consisting of three independent dimensions scored on a 7-point Likert scale.
  The emotional exhaustion (EE) scale, consisting of 9 items, identifies those individuals who are emotionally exhausted or overextended at work. The MBI has been extensively tested for reliability, validity, and internal consistency. Higher scores correspond to greater degrees of experienced burnout.
  Participants | 46 | 47 | 93
Maslach Burnout Inventory (MBI)-Depersonalization, % positive [Count of Participants; unit: Participants] — Maslach Burnout Inventory (MBI) is a 22-item self-report questionnaire consisting of three independent dimensions scored on a 7-point Likert scale.
  The depersonalization (DP) scale, consisting of 5 items, identifies those individuals who have an impersonal response towards recipients of their efforts. Higher scores correspond to greater degrees of experienced burnout.
  Participants | 41 | 37 | 78
Maslach Burnout Inventory (MBI)-Reduce Personal Accomplishment, % positive [Count of Participants; unit: Participants] — Maslach Burnout Inventory (MBI) is a 22-item self-report questionnaire consisting of three independent dimensions scored on a 7-point Likert scale.
  The personal accomplishment (PA) scale, consisting of 8 items, assesses lack of accomplishment and success related to work. Lower scores correspond to greater experienced burnout.
  Participants | 41 | 28 | 69

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Connor Davidson Resiliency Scale (CD-RISC) Scores
Description: The primary outcome is the pre-post changes in the CD-RISC scores in intervention and control subjects. The CD-RISC scale assesses resiliency in individuals. There are 25 items in the survey, each item is scored from 0-4, and the total ranges from 0-100. Higher scores indicate increased resiliency. Any individuals who score above 81 points on this survey will not qualify for this study as they are too inherently resilient. The study intervention will typically last 4 sessions, one session per week at a total of 4 weeks.
Time Frame: Once before the study intervention; one time immediately following the study intervention at 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 66.9 (9.1) | 67.6 (7.9)
  Post-Intervention | 73.6 (10.3) | 72.3 (9.4)

2. Secondary Outcome: Changes in Acceptability of the Sessions, on the Client Satisfaction Questionnaire (CSQ-8)
Description: This will be measured with the eight-item self-report Client Satisfaction Questionnaire (CSQ-8). This is survey has 8 items, and the total ranges from 1-32. Higher scores indicate higher satisfaction. The CSQ-8 will be administered before the intervention, weekly throughout the sessions and after the final treatment and control sessions.
Time Frame: Weekly during the 4 session/week intervention
Population: Some pts. did not complete the CSQ-8 survey each week, thus variations in the no. of participants analyzed each week for the MBCT cohorts exist.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 49 | 46
score on a scale
  Week 1 | 25.5 (3.1) | 26.2 (3.2)
  Week 2: number analyzed (Participants) | 48 | 40
  Week 2 | 25.4 (3.4) | 27.0 (3.0)
  Week 3: number analyzed (Participants) | 45 | 40
  Week 3 | 24.9 (4.4) | 28.2 (3.4)
  Week 4: number analyzed (Participants) | 42 | 37
  Week 4 | 25.5 (4.8) | 28.2 (3.8)

3. Secondary Outcome: Change From Baseline in Maslach Burnout Inventory (MBI) - Emotional Exhaustion Score
Description: Participants will also complete pre and post-intervention MBI surveys to assess changes in burnout symptoms. This survey is composed of 22 items. Each item is scored from 0-6. There are three questions domains: emotional exhaustion (9 items), depersonalization (5 items), and decreased person accomplishment (8 items). The items fall into one of these three categories and there are three domain scores. Higher values in each domain indicate increased burnout in that respective category.
  Scores for each item in the Emotional Exhaustion subscale are summed to obtain an overall score. Overall scores for the Emotional Exhaustion subscale can range between 0-54.
Time Frame: Once before the study intervention and once immediately after intervention at 4 weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 26.4 (9.8) | 29.2 (9.1)
  Post-Intervention | 24.9 (10.2) | 29.0 (9.1)

4. Secondary Outcome: Qualitative Interviews
Description: We will administer interviews to assess participant satisfaction with the intervention and control program. They will be administered to each group at the end of the intervention.
Time Frame: Once immediately after the study intervention at 4 weeks
Population: Data were not collected
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline in Post-traumatic Diagnostic Scale (PDS-5) - Intrusion Score
Description: Participants will complete pre/post-intervention PDS-5 surveys to assess post traumatic symptoms. This survey includes a pre-screen and 24 items. Each item is placed into the respective PTSD symptom category (as defined by the Diagnostic Statistical Manual-5) and scored. Higher scores in each symptom domain indicate increased chance of PTSD diagnosis. The domains are: intrusion (5 items), avoidance (2 items), changes in mood/cognition (7 items), and arousal/ hyperactivity (6 items). 2 items address "distress and interference" and 2 items address "symptom onset and duration.
  Scores for each question range from 0 to 3. The 5 items that contribute to the Intrusion score are summed to yield a possible range of PDS Intrusion scores of 0-15, with higher scores indicating greater intrusion.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 3.9 (3.1) | 4.3 (2.8)
  Post-Intervention | 3.7 (3.2) | 4.5 (3.2)

6. Secondary Outcome: Change From Baseline in HADS Anxiety Score
Description: Participants will also complete pre and post-intervention HADS surveys to assess changes in anxiety and depression symptoms. This survey has 14 items that fall into either the anxiety domain (7 items) or the depression domain (7 items). Items are scored 0-3 and scores, with higher scores indicating worse outcomes, and 11+ in each domain indicating abnormal cases.
  Scores for the 7 items in the anxiety domain are summed to yield a possible range of 0-21, with higher scores indicating more anxiety.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 9.6 (3.3) | 9.0 (3.4)
  Post-Intervention | 8.0 (3.2) | 8.6 (3.2)

7. Secondary Outcome: Changes From Baseline in the MBI-Depersonalization Score
Description: The Maslach Burnout Inventory (MBI) Depersonalization subscale is a 5-item self-report questionnaire that measures impersonal responses toward recipients of the respondent's efforts (e.g. patients). Scores can range between 0-30 with higher scores indicating greater depersonalization.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 10.8 (6.0) | 11.8 (5.7)
  Post-Intervention | 10.5 (6.5) | 12.7 (5.9)

8. Secondary Outcome: Change From Baseline in MBI- Personal Accomplishment Score
Description: The Maslach Burnout Inventory (MBI) Personal Accomplishment subscale is a 8-item self-report questionnaire that measures feelings of personal accomplishment and success related to work. Scores can range between 0-48 with higher scores indicating greater sense of accomplishment.
Time Frame: Once before the study intervention and once immediately after the 4 session intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 29.9 (6.3) | 30.8 (5.7)
  Post-Intervention | 34.1 (7.1) | 34.0 (6.5)

9. Secondary Outcome: Change From Baseline in PDS-5 Avoidance Score
Description: Participants will also complete pre/post-intervention PDS-5 surveys to assess post traumatic symptoms. This survey includes a pre-screen and 24 items. Each item is placed into the respective PTSD symptom category (as defined by the Diagnostic Statistical Manual-5) and scored. Higher scores in each symptom domain indicate increased chance of PTSD diagnosis. The domains are: intrusion (5 items), avoidance (2 items), changes in mood/cognition (7 items), and arousal/ hyperactivity (6 items). 2 items address "distress and interference" and 2 items address "symptom onset and duration.
  Scores for each question range from 0 to 3. The 2 items that contribute to the Avoidance score are summed to yield a possible range of PDS Avoidance scores of 0-6, with higher scores indicating greater avoidance.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 2.0 (1.6) | 1.9 (1.5)
  Post-Intervention | 1.5 (1.4) | 2.0 (1.7)

10. Secondary Outcome: Change From Baseline in PDS-5 Arousal Scores
Description: Participants will also complete pre/post-intervention PDS-5 surveys to assess post traumatic symptoms. This survey includes a pre-screen and 24 items. Each item is placed into the respective PTSD symptom category (as defined by the Diagnostic Statistical Manual-5) and scored. Higher scores in each symptom domain indicate increased chance of PTSD diagnosis. The domains are: intrusion (5 items), avoidance (2 items), changes in mood/cognition (7 items), and arousal/ hyperactivity (6 items). 2 items address "distress and interference" and 2 items address "symptom onset and duration.
  Scores for each question range from 0 to 3. The 6 items that contribute to the Arousal score are summed to yield a possible range of PDS Arousal scores of 0-18, with higher scores indicating greater arousal.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 5.1 (3.7) | 4.6 (3.5)
  Post-Intervention | 4.3 (4.3) | 5.0 (3.7)

11. Secondary Outcome: Change From Baseline in HADS-Depression Score
Description: Participants will also complete pre and post-intervention HADS surveys to assess changes in depression symptoms. This survey has 14 items that fall into either the anxiety domain (7 items) or the depression domain (7 items). Items are scored 0-3 and scores, with higher scores indicating worse outcomes, and 11+ in each domain indicating abnormal cases.
  Scores for the 7 items in the depression domain are summed to yield a possible range of 0-21, with higher scores indicating more depression.
Time Frame: Once before the study intervention and once immediately after the intervention at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Book Club Active Control | MBCT Intervention
Number analyzed (Participants) | 52 | 45
score on a scale
  Pre-intervention | 5.7 (4.0) | 5.8 (3.9)
  Post-Intervention | 4.5 (4.2) | 4.7 (4.1)

ADVERSE EVENTS:
Time Frame: Adverse Events were tracked for the duration of the study intervention, up to 4 weeks.
Arm/Group | Book Club Active Control | MBCT Intervention
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/58 | 0/48
Other Adverse Events (participants affected / at risk) | 0/58 | 0/48

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-13): https://cdn.clinicaltrials.gov/large-docs/20/NCT03132220/Prot_SAP_000.pdf